CLINICAL TRIAL: NCT04193995
Title: Intermittent Fasting as a Means to Lose Fluid Overload and Weight in Complicated Obesity: a Pilot Feasibility Study
Brief Title: Intermittent Fasting as a Means to Lose Fluid Overload and Weight in Complicated Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0460-18
Record Dates: First submitted 2019-09-15; First posted 2019-12-11 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2019-09

CONDITIONS: Intermittent Fasting; Obesity, Morbid; Comorbidities and Coexisting Conditions; Weight Loss; Fluid Retention
MeSH Terms: conditions — Intermittent Fasting; Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent fasting (Experimental): There are two 36h fasting periods (FP) every week, over a 12week period. Free access to water is allowed; two cups of tea or coffee are also allowed. Each 36h FP begins after the last meal, which is consumed no later than 2000h on the preceding nights. Fasting days are Sunday and Wednesday and fasting is terminated at 0800 on Monday and Thursday.
  Interventions: Behavioral: Intermittent fasting

INTERVENTIONS:
Behavioral: Intermittent fasting — There are two 36h fasting periods (FP) every week, over a 12week period. Free access to water is allowed; two cups of tea or coffee are also allowed. Each 36h FP begins after the last meal, which is consumed no later than 2000h on the preceding nights. Fasting days are Sunday and Wednesday, and fasting is terminated at 0800 on Monday and Thursday. Medications may be adjusted as needed during these visits, and this is reconsidered and may be further adjusted after the receipt of the blood tests results later during the day. Adjustments based on lab results are discussed with the patients during the clinic visit or later on the same day. Also, dietary needs are addressed by the physician and /or the dietician, during the clinic visit. As of week 3 through week 12, clinic visit is reduced to once a week, on Thursdays.

SUMMARY:
To examine the feasibility of intermittent fasting (36h, twice a week, unlimited salt and calorie-free fluid consumption), over three months, on body weight and composition in complicated obesity in whom age and medical complexity exclude the possibility of bariatric surgery.

DETAILED DESCRIPTION:
Rationale:

Complicated obesity: In weight loss-targeted treatment of obesity, current therapeutic choices include lifestyle modification, drug therapy, and bariatric surgery. For uncomplicated obesity, all the above comprise legitimate means. Attempted weight loss is traditionally initiated by targeting lifestyle, but unfortunately, the long term effect of this approach is limited as regards success rate, the extent of the achieved weight loss and the ability to sustain the achieved weight loss. The use of drugs is mostly reserved for cases where a limited weight loss of 5-10% is considered satisfactory. The safety of drug-assisted weight loss in older obese subjects with co-morbidities such as fluid retention, nephropathy, and heart failure remains insufficiently studied. Even for older subjects without such dominant conditions, data is scarce. For example, two trials (using phentermine/topiramate and liraglutide) have documented efficacy analyses between older adults and their younger, but enrolled only 7% (n= 5254) and 6.9% (n= 5232) older adults, respectively, among their study subjects. It is now well established that in non-elderly subjects, bariatric surgery is followed by substantial weight loss and leads to the cure of obesity and at least to a temporary amelioration/delay/cure of its sequels, including diabetes and hypertension.

However, weight loss is often most critically needed in subjects with complicated obesity, in whom an overall poor health state precludes bariatric surgery altogether. Individuals with long-standing obesity complicated by previous cardiovascular events, diabetes, renal impairment, fluid retention due to renal disease, the use of vasodilator drugs needed to control hypertension (alpha-blockers, calcium channel blocker), left ventricular diastolic dysfunction, respiratory dysfunction including obstructive sleep apnea, pulmonary hypertension, and restrictive lung disease. Such patients are generally too sick to be considered for bariatric surgery. In such patients concomitant weight loss from two body compartments could be extremely beneficial: reduction in fat mass and, often more critical in immediate terms, rapid loss of excess body fluids. In obesity complicated by clinically significant fluid retention, most of the excessive fluid volume is extra-vascular, residing in the extracellular tissue compartment, with only a small, though critical excess, occupying the intracellular compartment. Diuretics are the key tool to reduce volume overload, but they acutely lower the volume of the intravascular fluid compartment, which leads to impairment in renal, myocardial and general tissue arterial perfusion, thus often exacerbating renal failure and overall tissue hypoperfusion, including cerebral, myocardial and hepatic blood supply.

Most older and significantly obese subjects have had sustained obesity for several decades, which has allowed the cumulative evolution of at least some additional comorbidities such as the metabolic syndrome, diabetes, hyperlipidemia coronary heart disease, carotid artery stenosis and/or uncontrolled hypertension, congestive heart failure and renal disease. Paradoxically, then, those older subjects with a complex disease profile, who obviously comprise poor candidates for bariatric surgery, are also the group with the greatest immediate need to lose weight. It is therefore noteworthy that in Israel, individuals over the age of 65 cannot undergo bariatric surgery on the basis of obesity per se, unless approved by a special committee. Although European guidelines for the treatment of obesity in the elderly have concluded that the elderly should not be denied bariatric surgery solely on age grounds, long-term evidence in support of this statement is lacking such that both patients and physicians often consider bariatric surgery at this stage as too risky. Thus, current standard medical practice has little to offer to the complicated older obese patient who, on one hand is burdened with incapacitating obesity and its complications, and, on the other hand, is beyond the reach of the only tool to permanently alleviate obesity, i.e., bariatric surgery.

Intermittent and or short term fasting in humans: There is truly a lack of solid work on the safety and efficacy of fasting as a tool to lose weight in humans. The largest medical database on fasting has been collected on subjects practicing religious fast, such as the Ramadan. However, these forms of fasting are almost uniformly compensated for by excessive feeding either in the beginning or the end of the fast, or both. Insights on the effects of true fasting, longer than 24h, under medical supervision in humans is hard to find in published reports. In one study where caloric restriction for most of the week was combined with one day/week of nearly complete fasting (125Kcal), the intervention was deemed effective and unassociated with untoward effects in 54 obese women over a period of 24 weeks. A recent review included 16 studies of intermittent fasting in humans, of which 11 were carried out in overweight or obese subjects. Duration of the trials varied from 24h to 6 months. In two studies, fasting was daily and lasted from 11 and 16 hours within each day. There were 7 studies lasting 8-12 weeks, with alternate-day fasting, in which fasting was defined as consuming 20-30% of the required caloric intake on the fasting day. In two studies, caloric restriction was defined as consuming 25% less calories on the fasting day. As compared to a variety of more standard dietary measures, intermittent fasting appears to result in some modestly larger weight reduction. Among 16 intervention trials included in review, 11 reported statistically significant weight loss. However, in most of the reviewed intervention trials, complete fasting was either not attempted or restricted to 16 hours only, or less.

Complete intermittent fasting (excluding water) in humans: Despite the lack of data on the effects of complete intermittent fasting, however, a day of fasting is semi/non-intentionally practiced in many subjects undergoing investigative diagnostic procedures such as combined endoscopy and colonoscopy conducted in the afternoon or surgery unexpectedly postponed to the evening hours and many other medical conditions. Unfortunately, this unwanted form of fasting was never studied in depth. However, as early as the late 50s and early 60s of the previous century, it was noted that 5-7 days of complete fasting was associated with diuresis, natriuresis, and weight loss and appeared an effective mode of treatment of the failing heart, in otherwise treatment-refractory subjects who were, at that time, already "fully digitalized". An unexpected finding was the observation that water and salt excretion was enhanced during fasting: one of the fasting patients with heart failure lost 7.3 kg in 5 days, and the average daily weight loss of his 10 original subjects 0.85 kg to 1.5 kg per day, way above what might have been expected by the effect of negative caloric balance on fat and lean tissue loss alone.

Fasting diuresis and fasting as an ancillary tool to lower fluid overload Although it is well known that fasting in obese subjects is associated with natriuresis and development of cumulative negative sodium balance, the mechanism of increased urinary sodium excretion remains largely obscure. The leading hypothesis in recent decades was that reduction in insulin ameliorated increased insulin-driven re-absorption of sodium in the kidney, but overall, following the initial discovery of this phenomenon, it has attracted little research. It is also well established that the obese state, even uncomplicated by renal disease or congestive heart failure, is accompanied by a diminished ability to excrete salt.

During starvation, there appears to be an obligatory sodium loss in linkage to the metabolically generated organic anions, which further enhances fasting related natriuresis. Notably, unlike the action of diuretics and the tubular inhibition of sodium reabsorption, which lowers intravascular volume, the formation of organic anions during starvation takes place in the extravascular compartment, particularly in fat tissue, and would therefore allow the recruitment of tissue sodium (coupled to organic anions formed during lipolysis, and water), followed by the shift of sodium and water from the extravascular compartment to the intravascular compartment, and only then, excretion via the kidney. The latter process, therefore, does not lower intravascular fluid volume and should not impair renal perfusion and function. In support of this concept is the apparent dissociation between sodium and chloride excretion that has been reported with a relatively minimal increase in chloride excretion during the first week of fasting when sodium excretion is rapidly increasing. In fact, during the initial 3 days of fast in obese humans, natriuresis was proportional to urinary 3beta hydroxybutyrate excretion while urinary ammonium had not yet increased, thus indicating that the organic acids generated during lipolysis are the driving force in the shift of sodium from the body, outwards through the kidneys.

ELIGIBILITY:
Inclusion criteria 1)

1. Subjects with complicated obesity grade 2 or higher (Body Mass Index [BMI]>35kg/m2), i.e., obesity associated with renal failure with eGFR<60cc/min or heart failure with preserved ejection fraction (EF) (≥50%) and clinical evidence of fluid retention evidenced by the use of loop diuretic, or the presence of peripheral edema; or treatment in congestive heart failure clinics or history of admission to the hospital for heart failure during the past 3 years; OR • b. Subjects with complicated obesity, grade 2 or higher (BMI>35 kg/m2) [with renal failure as defined above-delete this requirement] and at least one of the following comorbidities: 1) Uncontrolled hypertension despite the use of at least 3 drugs administered at their maximal or close to maximal dose 2) Severe sleep apnea (based on a sleep lab report) 3) Pulmonary hypertension 4) Coronary heart disease 5) Type 2 diabetes mellitus 6) History of stroke (> 3 months prior to the recruitment to the trial) 2) Subjects who failed to lose weight on standard treatment, refuse standard medical treatment or are judged as unable to tolerate/unsuitable to receive standard medical treatment to lower body weight and in whom bariatric surgery is deemed unacceptable due to excessive surgical risk by the referring physician and/ or the PI and / or the patient and fulfill the following criteria

   1. Wish to fast 36 hours, twice a week, over three months
   2. Committed to attend the clinic at least once a week and perform blood tests every 2-14 days, as detailed in the protocol.
   3. Are well trained in-home glucose monitoring and are willing to monitor glucose levels during the fasting days.
   4. Are well trained in-home monitoring of blood pressure and are willing to measure blood pressure twice a day during the fasting days.
   5. Own and control a dependable means of 24/7 communication device, eg, cell phone, and are committed to avail this route of communication to the study staff.

Exclusion criteria:

1. Severe renal failure (eGFR<20cc/min)
2. Liver disease other than non-alcoholic fatty liver disease or cardiac cirrhosis or any liver disease with aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase levels>3 times of the upper limit of the normal range, albumin< 3.5 gr% or direct bilirubin>1.2 mg%.
3. Cognitive impairment assessed by a Mini-Mental State Exam (MMSE) score < 24
4. Living in a single household (caretaker is allowed)
5. Age less than 18 or >85 years
6. Pregnancy or intention to conceive or female at the reproductive age not using birth control means.
7. History of documented hypoglycemia during the past year despite attempted adjustment of treatment.
8. Unintended weight loss > 2kg over the past 2 months.
9. The initiation, within the study period of any one of the following medications, including topiramate, lyxumia, byetta, bydureon, belviq, Xenical, victoza, saxenda, trulicity, semaglutide or any other glucagon-like peptide-1 (GLP-1) analog. However, subjects already treated with these agents before the initiation of the trial may be included provided that the medication has been started at least 4 months prior to the beginning of the study and that weight loss during the 2 months preceding the trial did not exceed 2 kgs.
10. A subject who must use drugs whose use is not recommended on an empty stomach and in whom this qualification appears, in the investigator's opinion more critical than the potential chance to lose weight and excrete excess bodily fluids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Weight change | from baseline to 12 weeks
  % weight change
Fluid change | from baseline to 12 weeks
  % change in fluids (extracellular water as proxies for edema)
Fat percentage | from baseline to 12 weeks
  % change in fat percentage
Muscle mass | from baseline to 12 weeks
  % change in muscle mass

SECONDARY OUTCOMES:
Blood tests changes - glycemic control | from baseline to 12 weeks
  Fasting glucose (mg/dl)
Blood tests changes - glycemic control | from baseline to 12 weeks
  HbA1C (%)
Blood tests changes- lipid panel change | from baseline to 12 weeks
  Triglycerides, HDL and LDL cholesterol, total cholesterol) - change in mg/dl
Urine tests changes | from baseline to 12 weeks
  first urine void for creatinine, calcium, microalbumin, Na, K, Mg
Home sleep laboratory using watch PAT FDA-approved portable diagnostic device | from baseline to 12 weeks
  % change in % rapid eye movements (REM) of sleep time
Home sleep laboratory using WatchPAT™ FDA-approved portable diagnostic device | from baseline to 12 weeks
  % oxygen saturation change
24h ambulatory blood pressure monitoring (systolic and diastolic) | from baseline to 12 weeks
  % Systolic and diastolic change
Self-recorded diary ("recall 24"type) of caloric intake over 2 consecutive 24 hours is obtained | from baseline to 12 weeks
Fresh urine during visit to clinic for epigenetics | from baseline to 12 weeks
  The assessment of epigenetic variations, in the course of which the extracts undergo a bisulfite reaction do not allow genetic sequencing, and are directed to detect to identify areas of epigenetic changes without gene sequencing. Hence, no genetic information on the participating subjects will be obtained /recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Naftali Stern, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Institute of Endocrinology, Metabolism and Hypertension, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No